CLINICAL TRIAL: NCT05956535
Title: Air Optix® Night and Day® Aqua Therapeutic Wear
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: CLD265-N001
Record Dates: First submitted 2023-07-14; First posted 2023-07-21 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Bullous Keratopathy; Corneal Erosion; Entropion; Corneal Edema; Corneal Dystrophy
Keywords: Bandage lens
MeSH Terms: conditions — Entropion; Corneal Edema; Corneal Dystrophies, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- AONDA contact lenses: Lotrafilcon A contact lenses worn therapeutically as a bandage lens in a continuous wear (CW) modality (lenses worn continuously including overnight) as instructed by the eye care professional.
  Interventions: Device: Lotrafilcon A contact lenses
- PV2 contact lenses: Balafilcon A contact lenses worn therapeutically as a bandage lens in a continuous wear (CW) modality (lenses worn continuously including overnight) as instructed by the eye care professional.
  Interventions: Device: Balafilcon A contact lenses

INTERVENTIONS:
Device: Lotrafilcon A contact lenses — CE-marked silicone hydrogel contact lenses
  Other Names: Air Optix® Night and Day® Aqua; AONDA
  Groups: AONDA contact lenses
Device: Balafilcon A contact lenses — CE-marked silicone hydrogel contact lenses
  Other Names: PureVision® 2; PV2
  Groups: PV2 contact lenses

SUMMARY:
The purpose of this study is to support the safety and performance assessment of Air Optix Night and Day Aqua (AONDA) soft contact lenses for therapeutic use in accordance with updated EU Medical Device Regulation (MDR) requirements.

DETAILED DESCRIPTION:
In this retrospective, real world evidence study, the subjects wore Air Optix Night and Day Aqua (AONDA) soft contact lenses or PureVision 2 (PV2) soft contact lenses as a therapeutic lens for the treatment of a corneal condition with pain in one or both eyes as part of their eye care professional's treatment and management plan.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a corneal condition with pain for which AONDA or PV2 contact lenses were placed on one or both eye(s) as a therapeutic contact lens at Baseline.
* Baseline and Follow-up (up to 1 year from Baseline) charts available.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Had a condition (pathological, behavioral, and/or situational) that contraindicated therapeutic CL wear or confounds study results during the data collection period.
* Used systemic or ocular medication that would confound study results during the data collection period.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators will enroll charts following a pre-identified process.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline in corneal pain at the Follow-up Visit - Primary exposure | Baseline, Follow-up Visit (up to 1 year following the Baseline Visit)
  The Investigator will review the subject's chart and document change from baseline in corneal pain at the Follow-up visit as "improved, similar, or worsened." The Baseline Visit is defined as the first visit where the therapeutic contact lens was placed on eye as part of a treatment plan for a corneal condition. The Follow-up Visit is defined as the first visit where the therapeutic contact lens was removed from the eye, or the first visit following the removal of the contact lens if, for example, the contact lens was removed between visits. The primary exposure is defined as the first exposure to the study lens if, for example, there were multiple exposures to the study lens. The data collection period consists of any timeframe since and including 2009.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, CRD Vision Care, Study Director — Alcon Research, LLC
Locations (3):
- United States (3):
  - Delray Physician Care Center, Delray Beach, Florida
  - Koetting Associates, St Louis, Missouri
  - Contact Alcon Call Center For Trial Locations, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No